CLINICAL TRIAL: NCT07134244
Title: Development of Computational Models to Predict the Short-, Medium- and Long-term Cartilage Degeneration and Pain for Patients With Early-stage Osteoarthritis or Anterior Cruciate Ligament Injury
Acronym: MathKOA
Status: Recruiting | Type: Observational
Sponsor: Aalborg University (Other)
Collaborators: Lund University (Other); University of Eastern Finland (Other); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Morten Bilde Simonsen, Dr., Aalborg University
Other Study IDs: MathKOA_Cohort; NNF21OC0065373 (Other Grant/Funding Number: Novo Nordisk Fonden); N-20220057 (Registry Identifier: The North Denmark Region Committee on Health Research Ethics)
Record Dates: First submitted 2025-08-08; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee; Anterior Cruciate Ligament Injuries
Keywords: Knee joint; Cartilage degeneration; Biomechanics; Computational modeling; Pain assessment; Musculoskeletal modeling; Finite element analysis; MRI
MeSH Terms: conditions — Osteoarthritis, Knee; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Synovial fluid and blood samples will be collected from participants at designated study visits. These samples will be used for protein and biomarker analysis related to inflammation, cartilage metabolism, and disease progression. No DNA will be extracted or analyzed from any biospecimens. Samples will be stored under appropriate conditions until analysis is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Knee OA: Participants diagnosed with early-stage knee osteoarthritis. Followed longitudinally to assess cartilage degeneration, pain, and biomarkers.
- ACL reconstruction: Participants with a history of anterior cruciate ligament injury who have undergone reconstructive surgery. Monitored for cartilage health and OA progression.
- ACL No reconstruction: Participants with anterior cruciate ligament injury who did not undergo reconstructive surgery. Observed over time for cartilage degeneration and symptoms.
- Control for Knee OA group: Age- and sex-matched participants with no clinical or imaging signs of knee osteoarthritis. Serve as controls for the Knee OA group.
- Control for ACL reconstruction group: Participants with no history of ACL injury or surgery, matched to the ACL reconstruction group. Used as controls.
- Control for ACL No reconstruction group: Participants without knee injuries, matched to the ACL no reconstruction group. Serve as observational controls.

SUMMARY:
Knee osteoarthritis is a complex condition, and selecting effective non-drug treatments like orthoses or exercise is often difficult and imprecise. This study will follow individuals with early-stage knee osteoarthritis or previous anterior cruciate ligament injury to develop computational models that predict cartilage degeneration and pain over time. The models will integrate data from medical imaging, movement analysis, muscle strength testing, pain assessments, questionnaires, and biomarkers to improve personalized treatment planning.

ELIGIBILITY:
.3.1 ACL reconstruction group (n= 25) Inclusion criteria

* Adults under 70 years
* ACL injury within the last year and planned for ACL reconstruction at inclusion
* Informed consent form signed Exclusion criteria (at inclusion)
* Previous knee surgery before current knee trauma.
* Severe ischemic or neurological sequelae.
* BMI above 32.
* Clinically significant joint disease (inflammatory or degenerative) to other joints than the ACL injured knee (according to the clinician).
* Unsuitable for MRI (e.g. pacemaker or claustrophobia)
* Participants not able to fit the MRI knee coil (Thigh circumference larger than 73.5 cm measured 10 cm above the kneecap and a maximum calf circumferences of 61.5 cm).
* Drug addiction defined as the use of cannabis, opioids or other drugs as reported by the participant

ACL no reconstruction group (n= 25) Inclusion criteria

* Adults under 70 years
* ACL injury within the last year and with no plans for ACL reconstruction at inclusion
* Informed consent form signed Exclusion criteria (at inclusion)
* Previous knee surgery before current knee trauma.
* Severe ischemic or neurological sequelae.
* BMI above 32.
* Clinically significant joint disease (inflammatory or degenerative) to other joints than the ACL injured knee (according to the clinician).
* Unsuitable for MRI (e.g. pacemaker or claustrophobia)
* Participants not able to fit the MRI knee coil (Thigh circumference larger than 73.5 cm measured 10 cm above the kneecap and a maximum calf circumferences of 61.5 cm).
* Drug addiction defined as the use of cannabis, opioids or other drugs as reported by the participant

Early to moderate knee OA stage (n= 25) Inclusion criteria

* Adults under 70 years
* Diagnosis of knee OA (Kellgren Lawrence (KL) grade 1, 2 and 3 (Kohn et al., 2016). If there is no X-ray that is a maximum of 1 year old, a new one is taken.
* Stress-related pain in the knee and knee stiffness
* Informed consent form signed Exclusion criteria (at inclusion)
* Previous knee surgery
* Clinically significant joint disease (inflammatory or degenerative) of other joints than the knee at inclusion.
* Severe ischemic or neurological sequelae in the lower extremities.
* Clinically significant joint disease (inflammatory or degenerative) to other joints than the knees (according to the clinician).
* BMI above 32.
* Unsuitable for MRI (e.g., pacemaker or claustrophobia)
* Participants not able to fit the MRI knee coil (Thigh circumference larger than 73.5 cm measured 10 cm above the kneecap and a maximum calf circumferences of 61.5 cm).
* Drug addiction defined as the use of cannabis, opioids or other drugs as reported by the participant

Control groups (3 groups of 10 control participants matched for each of the patient groups, n=30) Inclusion criteria

* Adults under 70 years
* Informed consent form signed
* No radiological changes on a knee x-ray (Arendt-Nielsen et al., 2015). Exclusion criteria (at inclusion)
* Previous knee surgery
* Self-reported Knee problems (pain, stiffness)
* Clinically significant joint disease (inflammatory or degenerative) at inclusion.
* Severe ischemic or neurological sequelae in the lower extremities.
* BMI above 32.
* Unsuitable for MRI (e.g., pacemaker or claustrophobia)
* Participants not able to fit the MRI knee coil (Thigh circumference larger than 34.3-73.5 cm measured 10 cm above the kneecap and a maximum calf circumferences of 61.5 cm).
* Drug addiction defined as the use of cannabis, opioids, or other drugs as reported by the participant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Knee OA Participants diagnosed with early-stage knee osteoarthritis. Followed longitudinally to assess cartilage degeneration, pain, and biomarkers.
  ACL Reconstruction Participants with a history of anterior cruciate ligament injury who have undergone reconstructive surgery. Monitored for cartilage health and OA progression.
  ACL No Reconstruction Participants with anterior cruciate ligament injury who did not undergo reconstructive surgery. Observed over time for cartilage degeneration and symptoms.
  Control for Knee OA Group Age- and sex-matched participants with no clinical or imaging signs of knee osteoarthritis. Serve as controls for the Knee OA group.
  Control for ACL Reconstruction Group Participants with no history of ACL injury or surgery, matched to the ACL reconstruction group. Used as controls.
  Control for ACL No Reconstruction Group Participants without knee injuries, matched to the ACL no reconstruction group. Serve as observational controls.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2035-09-26 (Estimated); Study Completion 2036-09-26 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Cartilage Composition and Structure Assessed by Quantitative Magnetic Resonance Imaging | Data will be collected at three main time points: baseline, one-year follow-up, and three years follow-up. Additionally, a downscaled protocol will be used to follow the participants at 7- and 10 years follow-ups.
  Person-specific 3T MRI scans will be used to measure changes in knee cartilage, including T1ρ and T2 relaxation times and 3D geometry, as indicators of cartilage biochemical composition and structural integrity. Analyses will be used for predictive computational modeling of cartilage degeneration.

SECONDARY OUTCOMES:
Knee Pain Intensity (Visual Analog Scale) | Baseline, 1-year, 3-year, 7-year, 10-year follow-up.
  Self-reported knee pain intensity using a 100-mm Visual Analog Scale anchored with "0 = no pain" and "100 = worst imaginable pain.
Brief Pain Inventory Scores | Baseline, 1-year, 3-year, 7-year, 10-year follow-up.
  Severity and interference of pain over the past 24 hours, measured on a 0-10 scale using the Brief Pain Inventory questionnaire.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 1-year, 3-year, 7-year, 10-year follow-up.
  Self-administered questionnaire assessing pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. Scores range from 0 (no problems) to 4 (extreme problems) for each domain.
Hospital Anxiety and Depression Scale (HADS) - Total Score | Baseline, 1-year, 3-year, 7-year, 10-year.
  14-item self-report scale assessing anxiety and depression symptoms. Total score range: 0-42; higher scores indicate worse symptoms.
Pittsburgh Sleep Quality Index (PSQI) - Global Score | Baseline, 1-year, 3-year, 7-year, 10-year.
  19-item questionnaire assessing sleep quality over the past month. Global score range: 0-21; higher scores indicate poorer sleep quality.
Pain Catastrophizing Scale (PCS) - Total Score | Baseline, 1-year, 3-year, 7-year, 10-year.
  13-item scale assessing catastrophic thinking related to pain. Total score range: 0-52; higher scores indicate greater pain catastrophizing.
Short Form-12 Health Survey (SF-12) - Physical Component Summary (PCS) Score | Baseline, 1-year, 3-year, 7-year, 10-year.
  Summary measure of physical health-related quality of life. Score range: 0-100; higher scores indicate better physical health status.
Short Form-12 Health Survey (SF-12) - Mental Component Summary (MCS) Score | Baseline, 1-year, 3-year, 7-year, 10-year.
  Summary measure of mental health-related quality of life. Score range: 0-100; higher scores indicate better mental health status.
40-Meter Fast-Paced Walk Test - Time | Baseline, 1-year, 3-year.
  Time to walk 40 meters at fastest safe pace. Measured in seconds; lower scores indicate better performance.
30-Second Chair Stand Test - Number of Repetitions | Baseline, 1-year, 3-year.
  Number of full stands from a seated position completed in 30 seconds. Higher scores indicate better performance.
Stair Climb Test - Time | Baseline, 1-year, 3-year.
  Time taken to ascend a standard set of stairs. Measured in seconds; lower scores indicate better performance.
Timed Up-and-Go (TUG) Test - Time | Baseline, 1-year, 3-year.
  Time to rise from a chair, walk 3 meters, turn, return, and sit. Measured in seconds; lower scores indicate better performance.
3D Motion Capture - Kinematic Parameters | Baseline, 1-year, 3-year.
  Joint angles and Movements patterns during movement, measured in degrees, using 3D motion capture.
3D Motion Capture - Kinetics Parameters | Baseline, 1-year, 3-year.
  Inverse dynamics calculated from movement patterns and force plates during activities, using 3D motion capture.
Motion capture Surface Electromyography (EMG) | Baseline, 1-year, 3-year.
  Muscle activation amplitude from selected lower limb muscles, measured in microvolts (µV) and processed per SENIAM guidelines.
Pressure Pain Detection Threshold | Baseline, 1-year, 3-year.
  Minimum pressure at which a sensation becomes painful, measured in kilopascals (kPa) using a computer-controlled cuff algometer. Higher values indicate reduced sensitivity to pain.
Pressure Pain Tolerance Threshold | Baseline, 1-year, 3-year.
  Maximum pressure a participant can tolerate, measured in kilopascals (kPa). Higher values indicate greater pain tolerance.
Temporal Summation of Pain | Baseline, 1-year, 3-year.
  Increase in pain intensity in response to repetitive stimulation, measured as change in pain rating on a 0-10 numeric rating scale. Higher scores indicate greater central sensitization.
Conditioned Pain Modulation Effect | Baseline, 1-year, 3-year.
  Percentage change in pain rating during a conditioning stimulus, indicating efficiency of endogenous pain inhibition. Higher percentages indicate stronger pain inhibition.
Plasma Protein Biomarker Concentrations - Inflammatory Markers | Baseline, 1-year, 3-year, 7-year, 10-year.
  Quantitative concentrations of inflammatory biomarkers in plasma using LC-MS/MS and high-multiplex immunoassays (Olink). Higher or lower values indicate changes in inflammatory status.
Plasma Protein Biomarker Concentrations - Cartilage Metabolism Markers | Baseline, 1-year, 3-year, 7-year, 10-year.
  Quantitative concentrations of cartilage metabolism biomarkers in plasma. Higher or lower values indicate changes in cartilage turnover.
Synovial Fluid Protein Biomarker Concentrations - Inflammatory Marker | Baseline, 1-year, 3-year, 7-year, 10-year.
  Quantitative concentrations of inflammatory biomarkers in synovial fluid
Synovial Fluid Protein Biomarker Concentrations - Cartilage Metabolism Markers | Baseline, 1-year, 3-year, 7-year, 10-year.
  Quantitative concentrations of cartilage metabolism biomarkers in synovial fluid

CONTACTS AND LOCATIONS:
Overall Officials: Michal Skipper Andersen, Phd, Principal Investigator — Department of Materials and Production, Aalborg University, Denmark
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg, North Denmark
  - Aalborg University, Aalborg, Northen Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Undecided